CLINICAL TRIAL: NCT07040085
Title: Effects of Y-6 Sublingual Tablets for Patients With Acute Ischemic Stroke: a Randomised, Double-blind, Multicenter, Placebo-controlled Phase 3 Trial (FUTURE-2)
Brief Title: Y-6 Sublingual Tablets for Patients With Acute Ischemic Stroke
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Beijing Tiantan Hospital (Other)
Collaborators: Neurodawn Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Principal Investigator, yilong Wang, PI，chief physician, Beijing Tiantan Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: YW2025-020-01
Record Dates: First submitted 2025-06-10; First posted 2025-06-26 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-05

CONDITIONS: Stroke
Keywords: Y-6; stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Y-6 (Experimental): Take the Y-6 sublingual tablet (each tablet contains 6 mg Dexborneol and 25 mg Cilostazol ), for 28 days continuously.
  Interventions: Drug: Y-6
- Y-6 placebo (Placebo Comparator): Take the placebo of Y-6 sublingual tablet (each tablet contains 0.06 mg Dexborneol and 0 mg Cilostazol ), for 28 days continuously.
  Interventions: Drug: Y-6 placebo

INTERVENTIONS:
Drug: Y-6 — each tablet of Y-6 contained 6 mg of dexborneol and 25 mg of cilostazol; Both groups took one tablet q12h for 28 days.
  Arms: Y-6
Drug: Y-6 placebo — each tablet of Y-6 placebo contained 0.06 mg of dexborneol and 0 mg of cilostazol. Both groups took one tablet q12h for 28 days.
  Arms: Y-6 placebo

SUMMARY:
This study aims to evaluate the efficacy of Y-6 sublingual tablets in improving microcirculation dysfunction and reducing thrombo-inflammation in patients who had AIS caused by LVO and will receive EVT. Moreover, we expect to evaluate the safety of using Y-6 sublingual tablet in such study population.

This study rationale is based on the following scheme: in patients with acute ischemic stroke caused by LVO, receiving reperfusion therapy may cause futile recanalization and thus lead to microcirculation dysfunction and thrombo-inflammation as consequences. Dexborneol has anti-inflammatory effects and Cilostazol has antiplatelet effects and BBB protection; therefore, the multi-component tablet may exert neuroprotective effects in terms of improving microcirculation dysfunction and reducing thrombo-inflammation in patients with AIS after reperfusion therapy.

The primary purpose of this study is to investigate the proportion of modified-Rankin scale (mRS) score recovered to 0~1 score at 90 days after randomization.

The follow-up duration is 3 months, and the visit schedule is as follows: Subjects enrolled based on randomization procedures will receive visits at screening/baseline period, 1 day, 7 days, 28 days and 90 days after randomization, and in case of any events.

ELIGIBILITY:
Inclusion Criteria:

* 35 years old ≤ Age ≤ 80 years old;
* Patients with acute ischemic stroke diagnosed within 24 hours of onset (time from onset to start of endovascular treatment);
* Patients with first stroke or mRS score 0-1 prior to this onset ;
* Patients with acute intracranial large vessel occlusion (LVO) confirmed by imaging examination, including occlusion of intracranial segments of internal carotid arteries, T-shaped bifurcation, MCA M1 and/or M2 segments and ACA A1 and/or A2 segments;
* ASPECTS score ≥ 6 at screening;
* 6<NIHSS score ≤ 25 after this onset;
* Patients who had the indications for endovascular treatment and were scheduled for endovascular treatment;
* Patients or his/her legal representatives were able to understand and sign the informed consent.

Exclusion Criteria:

* Patients who are allergic to the active ingredients or excipients of investigational products；
* Severe disorder of consciousness at screening: NIHSS 1a consciousness level ≥2 points;
* Patients with previously diagnosed intracranial haemorrhage at screening, including parenchymal hemorrhage, intraventricular hemorrhage, subarachnoid hemorrhage, subdural/external hematoma, etc.;
* Patients with previously diagnosed intracranial tumor, arteriovenous malformation, or aneurysm at screening;
* Patients with previously diagnosed congestive heart failure at screening;
* Patients with bilateral LVO at anterior circulation or LVO at posterior circulation or LVO of unknown aetiology at screening;
* Patients who have received treatment with warfarin, novel oral anticoagulants, argatroban, snake venom, defibrase, lumbrokinase and batroxobin after onset;
* Patients with severe hematologic abnormality or severe hepatic insufficiency or renal insufficiency and received dialysis for various reasons at screening (hematologic abnormality was defined as platelet count <100×109/L; severe hepatic insufficiency was defined as ALT > 3 × ULN or AST >3 × ULN; severe renal insufficiency was defined as serum creatinine >3.0 mg/dl (265.2 μmol/L) or creatinine clearance < 30 ml/min);
* Patients with previously diagnosed hemorrhagic tendency (including but not limited to): hemorrhagic retinopathy or hereditary hemorrhagic disorders, such as hemophilia, at screening;
* Patients with refractory hypertension that is difficult to be controlled by medication (systolic blood pressure > 180 mmHg or diastolic blood pressure > 110 mmHg);
* Patients with history of major head trauma or stroke within 1 month prior to randomization;
* Patients who have received intracranial or spinal surgery within 3 months prior to randomization;
* Patients with history of major surgery or serious physical trauma within 1 month prior to randomization;
* Male subjects (or their mates) or female subjects who had planned to have a child during the whole study period and within 3 months after the end of the study period or were unwilling to use one or more non-drug contraceptive methods (e.g., complete abstinence, condoms, ligation, etc.) during the study period;
* Patients with contraindications to known contrast agents or other contrast agents;
* Patients who plan to receive other surgical or intervention therapy within 3 months, which might require discontinuation of the study drugs;
* Patients with life expectancy of less than 3 months;
* Patients who have received treatment of investigational drugs or devices within previous 3 months;
* Other investigator-evaluated conditions which may influence the compliance of patients or where it is not suitable for patients to participate in this trial.

Ages: 35 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 892 (Estimated)
Dates: Start 2025-08-05 (Estimated); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Proportion of subjects whose mRS recover to 0-1 at 90 days after randomization. | 90 days
  mRS recover to 0-1

SECONDARY OUTCOMES:
•mRS at 90 days after randomization | 90 days
  mRS (0-6); the scale ranges from 0 to 5, where 0 indicates no symptoms, and 5 signifies severe disability requiring continuous care and assistance. 6, denotes death.
• Changes in NIHSS from baseline to 1 day, 7 days and 28 days after randomization； | from baseline to 1 day, 7 days and 28 days
  Changes in NIHSS; the total score ranges from 0 to 42, with lower scores indicating better neurological status.
• Proportion of patients with early neurological deterioration at 1 day after randomization; | at 1 day
  early neurological deterioration
• Proportion of subjects with combined vascular events at 90 days after randomization. | 90 days
  combined vascular events

OTHER OUTCOMES:
• Incidence and severity of treatment emergent adverse events (TEAEs) across treatment groups | During the 90 days
  TEAEs
• Changes in laboratory test results after treatment; | During the 90 days
  Changes in laboratory test results (such as the red blood cell count, white blood cell count, platelets, blood biochemical indicators, etc.. )
• Changes in vital signs after treatment | During the 90 days
  • Changes in vital signs after treatment（ including blood pressure, pulse, breathing, and other indicators.）
• Changes in physical examination findings after treatment | During the 90 days
  • Changes in physical examination findings after treatment: Lungs, Gastrointestinal tract, Urinary system, Musculoskeletal system, Skin, Lymph nodes, et
• Incidence of symptomatic intracranial haemorrhage at 28 days after treatment (per Heidelberg heamorrhage classification) | at 28 days
  Symptomatic intracranial haemorrhage Heidelberg heamorrhage classification
• Incidence of any bleeding events after treatment | During the 90 days
  • Incidence of any bleeding events after treatment
• Incidence of vascular deaths； | During the 90 days
  • Incidence of vascular deaths；
• Incidence of all-cause deaths after treatment | During the 90 days
  • Incidence of all-cause deaths after treatment
• Incidence of platelet count ≤100×10^9/L after treatment | During the 90 days
  • Incidence of platelet count ≤100×10^9/L after treatment

IPD SHARING:
Plan to Share IPD: No